CLINICAL TRIAL: NCT05699213
Title: A Pilot Study Evaluating the Feasibility of Novel MRI Sequences and Blood-Based Biomarkers for Discriminating Nodules Found During Lung Cancer Screening
Brief Title: MRI and Biomarkers for Lung Nodules Detected During Lung Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Sara Ghandehari, Associate Professor, Cedars-Sinai Medical Center
Other Study IDs: STUDY00002249
Record Dates: First submitted 2022-12-09; First posted 2023-01-26 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: Lung MRI — MRI of the lung
Diagnostic Test: Blood Draw — Blood Draw

SUMMARY:
The primary objective of this pilot observational study is to evaluate the accrual and retention rate of a study population from a centralized lung cancer screening program to support MRI and blood-based biomarker research for lung cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and understand informed consent
* Male or female adults who are at high risk for lung cancer and are enrolled in the centralized lung cancer screening program: Based on USPSTF guidelines: Age 50-80 with 20 or greater pack-year smoking story who continue to smoke or quit within the past 15 years without sign or symptoms of lung cancer. Or based on National Comprehensive Cancer Network (NCCN) guidelines but do not meet the USPSTF guidelines, age 50-unlimited
* Found to have one or more lung nodules that is 6mm or greater on screening LDCT

Exclusion Criteria:

* Persons with an active diagnosis of cancer
* Persons with active signs or symptoms of lung cancer
* Persons with mechanically, magnetically, or electrically activated implants, such as cardiac pacemakers, neurostimulators, and infusion pumps.
* Persons with ferromagnetic implants and ferromagnetic foreign bodies, such as intracranial aneurysm clips, shrapnel and intraocular metal chips as these could become dislodged.
* Persons who are pregnant, nursing, are implanted with intrauterine devices (IUD's) that are not MR-compatible
* Persons unable to tolerate MRI imaging secondary to an inability to lie supine or severe claustrophobia.
* Persons who are non-compliant with visit instructions, including inability to lie still, hold breath or follow procedure instructions

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The primary subject population will be patients who qualify for lung cancer screening based on United States Preventive Services Taskforce (USPSTF) guidelines: Age 50-80 with 20 or greater pack-year smoking history who continue to smoke or have quit within the past 15 years without sign or symptoms of lung cancer.
  The secondary subject population will be patients who are at increased risk of lung cancer based on National Comprehensive Cancer Network (NCCN) guidelines, but do not meet the USPSTF guidelines
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Accrual and Retention Rate | 3 years
  The primary outcome measure is the accrual and retention rate of a study population from a centralized lung cancer screening program to support MRI and blood-based biomarker research.

SECONDARY OUTCOMES:
Concordance of Size of Nodules | 3 Years
  The secondary objective of this study is to evaluate the concordance of imaging features of nodules on LDCT versus MRI in a screening population. Concordance of the size of nodules on LDCT versus MRI will be analyzed using Bland Altman and linear regression.
Concordance of Nodule Features: Presence of Calcifications | 3 years
  The secondary objective of this study is to evaluate the concordance of imaging features of nodules on LDCT versus MRI in a screening population. Concordance for the presence of calcifications will be analyzed using McNemar's test, sensitivity and specificity.
Concordance of Nodule Features: Presence of Fat | 3 years
  The secondary objective of this study is to evaluate the concordance of imaging features of nodules on LDCT versus MRI in a screening population. Concordance for the presence of fat will be analyzed using McNemar's test, sensitivity and specificity.
Concordance of Nodule Features: Presence of Spiculations | 3 years
  The secondary objective of this study is to evaluate the concordance of imaging features of nodules on LDCT versus MRI in a screening population. Concordance for the presence of spiculations will be analyzed using McNemar's test, sensitivity and specificity.
Concordance of Nodule Features: Solid, Part Solid, Non-Solid | 3 years
  The secondary objective of this study is to evaluate the concordance of imaging features of nodules on LDCT versus MRI in a screening population. Concordance for whether the nodule is solid, part solid, or non-solid will be analyzed using McNemar's test, sensitivity and specificity.

OTHER OUTCOMES:
Exploratory Outcomes | 3 years
  The exploratory objectives of this study are to generate preliminary data in support of larger studies in a lung cancer screening population looking at: 1) the use of genetic biomarkers and 2) the use of novel MRI acquisition parameters and radiomics

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ghandehari, MD, Principal Investigator — Cedars-Sinai
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States